CLINICAL TRIAL: NCT02607007
Title: The Effect of Dairy and Non-dairy Breakfasts on Subjective Appetite Ratings, Food Intake, and Post-meal Glycemia in Healthy Older Adults
Brief Title: The Effect of Dairy and Non-dairy Breakfasts on Satiety and Post-meal Glycemia in Healthy Older Adults
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Toronto (Other)
Collaborators: Dairy Farmers of Canada (Other)
Responsible Party: Principal Investigator, G. Harvey Anderson, Professor, University of Toronto
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: DFC_31936
Record Dates: First submitted 2015-11-13; First posted 2015-11-17 (Estimated); Last update posted 2016-05-12 (Estimated); Status verified 2016-05

CONDITIONS: Diabetes; Obesity
Keywords: Dairy; Post-prandial Glycemia; Satiety; Food Intake; Insulin; Milk; Greek yogurt; Cheese; Soy beverage
MeSH Terms: conditions — Diabetes Mellitus; Obesity; Insulin Resistance | interventions — Milk; Yogurt; Soy Milk; Water

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- 2% M.F. Milk (Experimental): Breakfast meal: 250 mL 2% M.F. milk, 75 g white toast, 23.2 g strawberry jam, 100 mL water
  Interventions: Other: 2% M.F. Milk; Other: White Bread; Other: Strawberry Jam
- 2% M.F. Plain Greek Yogurt (Experimental): Breakfast meal: 175 g 2% plain Greek yogurt, 75 g white toast, 23.2 g strawberry jam, 100 mL + 75 mL water
  Interventions: Other: White Bread; Other: Strawberry Jam; Other: 2% M.F. Plain Greek yogurt
- 31% M.F. Cheddar Cheese (Experimental): Breakfast meal: 30 g 31% M.F. cheddar cheese, 75 g white toast, 27.0 g strawberry jam, 100 mL + 220 mL water
  Interventions: Other: White Bread; Other: Strawberry Jam; Other: 31% M.F. Cheddar Cheese
- Soy Beverage (Experimental): Breakfast meal: 250 mL soy beverage, 75 g white toast, 19.3 g strawberry jam, 100 mL water
  Interventions: Other: White Bread; Other: Strawberry Jam; Other: Soy Beverage
- Water (control) (Experimental): Breakfast meal: 250 mL + 100 mL water
  Interventions: Other: Water

INTERVENTIONS:
Other: 2% M.F. Milk
  Other Names: 2% cow's milk; Neilsen Canada; White milk
  Arms: 2% M.F. Milk
Other: White Bread
  Other Names: White toast; Wonder Bread Canada
  Arms: 2% M.F. Milk; 2% M.F. Plain Greek Yogurt; 31% M.F. Cheddar Cheese; Soy Beverage
Other: Strawberry Jam
  Other Names: Pure strawberry jam (not seedless); Fruit jam; Smucker's
  Arms: 2% M.F. Milk; 2% M.F. Plain Greek Yogurt; 31% M.F. Cheddar Cheese; Soy Beverage
Other: 31% M.F. Cheddar Cheese
  Other Names: Mild cheddar cheese; Hard cheese; Armstrong Canada
  Arms: 31% M.F. Cheddar Cheese
Other: 2% M.F. Plain Greek yogurt
  Other Names: Yogurt; Oikos, Danone Canada
  Arms: 2% M.F. Plain Greek Yogurt
Other: Soy Beverage
  Other Names: Soy milk; Non-dairy alternative; So Good, Vanilla
  Arms: Soy Beverage
Other: Water
  Other Names: Calorie-free control
  Arms: Water (control)

SUMMARY:
This study investigates the effects of dairy breakfasts (2% cow's milk, 2% Greek yogurt, cheese) and a non-dairy breakfast (soy beverage) on satiety and post-meal blood glucose. Each participant will receive every treatment in this crossover design study.

DETAILED DESCRIPTION:
Regular consumption of dairy is associated with better body composition and lower incidences of type 2 diabetes and obesity. This may be due to dairy's ability to increase satiety and decrease post-prandial glycemia. However, most clinical studies have only investigated isolated dairy proteins (whey and casein) and the effects of whole dairy products, consumed as part of a meal, remain unclear. Additionally, the effect of dairy type and form remain to be further investigated. Therefore, this study will test the effects of dairy products when consumed with a high glycemic index breakfast on satiety and post-prandial glycemia.

Thirty healthy older males and females (60-70 years, BMI 18.5-30.0 kg/m2) will be recruited for the randomized, unblinded, crossover study. Participants will fast overnight, and at baseline will consume 1) 2% milk (250 mL), 2) soy beverage (250 mL), 3) plain 2% Greek yogurt (175 g), 4) cheddar cheese (30 g), or 5) water (250 mL - control). Treatments will be consumed along with 2 pieces of white toast with strawberry jam, except for the water control which will be consumed alone. All breakfast meals will be isocaloric and water will be given with the yogurt (75 mL) and cheese (220 mL) to compensate for fluid content. At 0 (baseline), 15, 30, 45, 60, 90, 120, 150, 180, (pre-meal period) and 210 minutes (post-meal period) blood will be collected for glucose analysis and subjective appetite ratings completed. Insulin will be analyzed every 30 minutes. Between 180-200 minutes, an ad libitum lunch will be provided to assess food intake.

ELIGIBILITY:
Inclusion Criteria:

* Healthy BMI (18.5-30.0 kg/m2)
* Regular breakfast consumers
* Menopausal for at least 1 year (females)

Exclusion Criteria:

* Smoking
* Diabetes
* Fasting blood glucose equal to or higher than 6.0 mmol/L
* Cardiovascular disease
* Medication affecting appetite or metabolism
* Trying to lose or gain weight through a diet or exercise regime
* Lactose intolerance or allergies to study foods
* Score equal to or higher than 11 on Eating Habits Questionnaire

Ages: 60 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2015-10; Primary Completion 2015-12 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Blood Glucose | 0-210 minutes
  Blood glucose (mmol/L) is measured using finger prick capillary blood samples
Subjective Appetite | 0-210 minutes
  Subjective appetite ratings are obtained from four 100 mm visual analogue scale (VAS) questions assessing "Desire to Eat", "Hunger", "Fullness" and "Prospective Food Consumption". The average of all four VAS is calculated to obtain the average appetite score for statistical analysis.

SECONDARY OUTCOMES:
Insulin | 0-210 minutes
  Blood insulin (μU/mL) is measured using finger prick capillary blood samples
Food Intake | 180-200 minutes
  Food at an ad libitum lunch meal consisting of a dish of rice, meatballs, and tomato sauce will be weighed to determine food intake based on nutrition information provided by the manufacturers.

CONTACTS AND LOCATIONS:
Overall Officials: G. Harvey Anderson, Ph.D., Principal Investigator — Department of Nutritional Sciences, University of Toronto
Locations (1):
- Department of Nutritional Sciences, University of Toronto, Toronto, Ontario, Canada